CLINICAL TRIAL: NCT01564147
Title: More Added Value of Therapeutic Education in the Management of Patients With Rheumatoid Arthritis
Brief Title: More Added Value of Therapeutic Education in the Management of Patients With Rheumatoid Arthritis (ETP-PR)
Acronym: ETP-PR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BRD/11/02-J
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Therapeutic Education, Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Education therapeutic (Other): Access to the course of immediate therapeutic education
  Interventions: Other: immediate therapeutic education
- therapeutic education delayed (Other): Group receiving therapeutic education 6 months later (control group)
  Interventions: Other: therapeutic education delayed

INTERVENTIONS:
Other: immediate therapeutic education — Access to the course of immediate therapeutic education
  Arms: Immediate Education therapeutic
Other: therapeutic education delayed — Group receiving therapeutic education 6 months later (control group)
  Arms: therapeutic education delayed

SUMMARY:
Taking into account the recommendations of the Health Authority [1] and the application of patients' associations, we have structured a course of therapeutic education includes three stages for patients with rheumatoid arthritis and followed at Nantes University Hospital. Step 1: initial interview with a nurse patient education for diagnosis and education with the patient to choose three subjects from among 10 offered him problematic; Step 2: Orientation in an educational path that provides access to 6 months group workshops (3 maximum) and / or interviews tailored to the three selected topics; Step 3: final interview with a nurse said therapeutic education formative assessment to take stock. The main objective of our work is to ensure that the patient finds it easier solutions to the three problematic topics him after 6 months of education after six months without treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting at clinics for Rheumatology or the Rheumatology Day Hospital at the University Hospital or hospitalized in the department of Rheumatology
* Men or women
* Having signed the consent
* major
* Affiliated to social security or covered by the CMU
* Patient with rheumatoid arthritis meeting the ACR criteria
* Patient with rheumatoid arthritis stable for at least 6 months (change in DAS 28 <1.2)

Exclusion Criteria:

* Patient can not understand the information
* Patient confined to bed or chair, unable to care for himself or not doing with difficulty
* pregnant patient
* minors
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
EVA measures the overall ability to find solutions applicable to their situation | 12 months
  Investigate whether, overall, the patient is more easily applicable solutions to the situation after six months of therapeutic education after six months without therapeutic education for three problems identified after the initial filling of the questionnaire (controls ) and after the initial interview with the nurse (test group)

SECONDARY OUTCOMES:
EVA measures the ability to find solutions applicable to their situation for each of the three problems identified. | 12 months
  Ability to find solutions applicable to their situation for each of the three problems identified
Knowledge (score / 10) treatments for rheumatoid arthritis, knowledge (note/10) signs of a flare of rheumatoid arthritis. | 12 months
  Skills that we consider indispensable
Self-efficacy against a disease flare (EVA), self-efficacy against a side effect of treatment (EVA) | 12 months
  Perceived self-efficacy compared to rheumatoid arthritis
RAPID score 4 (scale) | 12 months
  Scalability of rheumatoid arthritis
EVA measuring fatigue | 12 months
  Fatigue
Duration of morning stiffness in minutes or hours. | 12 months
  Duration of stiffness
CRP and VS | 12 months
  Biological criteria
Scale of STAI S Scale of STAI S | 12 months
  Anxiety
Beck Scale | 12 months
  Depression
Evaluation Test of adherence of Girerd | 12 months
  Observance
Dosage Cortancyl or Solupred. | 12 months
  Use of steroids
Number of visits to physician, rheumatologist at at therapist, psychiatrist, occupational physician, number of hospitalizations, number of meetings with occupational therapist, social worker, dietician, physiotherapist, psychologist... | 12 months
  Consumption of medical and paramedical
Patient satisfaction with respect to information received, the caller and the improvement in different areas of health (EVA) | 12 months
  Satisfaction with patient education
Attendance at meetings / workshops offered after the initial diagnosis. | 12 months
  Membership

CONTACTS AND LOCATIONS:
Overall Officials: Yves Maugars, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Maugars, Nantes, France